CLINICAL TRIAL: NCT00006110
Title: Nonrandomized Ph II Study of Multimodality Therapy for Stg IIB, IIIA/B, or Stg IV Breast Cancer w/4 Cycles of Adriamycin and Cytoxan (AC),Followed by 12 Weeks of Paclitaxel w/ or w/o Herceptin Followed by Local Therapy Followed by Wkly Herceptin or no Additional Therapy
Brief Title: Multimodality Treatment for Women With Stage II, Stage III, or Stage IV Breast Cancer
Acronym: NRR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 9818; LCCC9818 (Other: UNC Lineberger Comprehensive Cancer Center); NCI-G00-1836 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Trastuzumab; Cyclophosphamide; Doxorubicin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neo-adjuvant Herceptin with or without radiation (Experimental): Chemotherapy followed by Taxol plus Herceptin followed by surgery followed by radiation (or no radiation) followed by additional Herceptin
  Interventions: Biological: trastuzumab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel; Procedure: conventional surgery
- Non-Herceptin with or without radiation (Experimental): Chemotherapy followed by Taxol followed by surgery followed by radiation (or no radiation)
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel; Procedure: conventional surgery

INTERVENTIONS:
Biological: trastuzumab — infusion 4 mg/kg load week 1; 2 mg/kg weekly thereafter for 12 weeks
  Other Names: Herceptin
  Arms: Neo-adjuvant Herceptin with or without radiation
Drug: cyclophosphamide — 600 mg/m2, intravenous infusion every 3 weeks for four cycles
  Other Names: Lyophilized Cytoxan; Endoxan; Cytoxan; Neosar; Procytox; Revimmune; Cycloblastin
Drug: doxorubicin hydrochloride — 60 mg/m2 intravenously, 5-10 minutes, every 3 weeks, up to 12 weeks
  Other Names: Adriamycin
Drug: paclitaxel — 90 mg/m2 weekly, intravenously 1 hour after herceptin, given weekly up to 12 weeks or 175 mg/m2, intravenously every 3 weeks, up to 12 weeks (only if not receiving Herceptin®)
  Other Names: Taxol
Procedure: conventional surgery — Surgical excision will take place 12-13 weeks for the neo-adjuvant herceptin setting and 12-13 weeks in the non-herceptin setting. Surgery will take place prior to chemotherapy in the adjuvant herceptin setting

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining chemotherapy, monoclonal antibody therapy, and surgery may be a more effective treatment for breast cancer.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy, monoclonal antibody therapy, and surgery in treating women who have stage II, stage III, or stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the cardiac and other toxicity of paclitaxel when administered with trastuzumab (Herceptin) after doxorubicin and cyclophosphamide in women with stage IIB, IIIA, IIIB, IIIC, or previously untreated stage IV breast cancer.
* Determine whether the addition of paclitaxel with or without trastuzumab to conventional breast cancer adjuvant therapy (doxorubicin and cyclophosphamide) further decreases tumor size and the number of positive axillary nodes in these patients.
* Determine the 5-year disease-free survival and overall survival of patients treated with these regimens.
* Determine whether the initial pathologic response in patients receiving neoadjuvant therapy correlates with the eventual 5-year disease-free survival or overall survival.
* Compare the number of patients eligible for breast-conserving cancer surgery after treatment with doxorubicin and cyclophosphamide vs paclitaxel and trastuzumab.
* Correlate clinical and radiographic response rate with pathologic response rate in the primary tumor and axillary lymph nodes and determine which parameter best determines the pathologic response rate in patients treated with these regimens.

OUTLINE: Patients either received neoadjuvant therapy (HER-2 overexpressing and non-overexpressing patients) or adjuvant therapy (HER-2 overexpressing patients only).

* Neoadjuvant therapy: Patients receive one of two treatment regimens.

  * Regimen I (HER-2 non-overexpressing patients or HER-2 overexpressing patients who refuse trastuzumab (Herceptin) therapy): Patients receive doxorubicin IV and cyclophosphamide IV over 30 minutes and paclitaxel IV over 3 hours on day 1 every 3 weeks for a total of 4 courses. Patients then undergo surgery with or without adjuvant radiotherapy and/or oral tamoxifen.
  * Regimen II (HER-2 overexpressing patients only): Patients receive doxorubicin and cyclophosphamide as in regimen I. After completion of course 4, patients receive paclitaxel IV and trastuzumab IV over 90-150 minutes weekly on weeks 13-24. Patients then undergo surgery with or without adjuvant radiotherapy. Patients then receive trastuzumab IV over 30 minutes weekly on weeks 29-69 if they did not receive radiotherapy or on weeks 36-76 if they did receive radiotherapy.
* Adjuvant therapy: Patients who receive adjuvant therapy (HER-2 overexpressing patients only) receive doxorubicin IV and cyclophosphamide IV over 30 minutes on day 1 every 3 weeks for a total of 4 courses. After completion of course 4, patients receive paclitaxel IV and trastuzumab IV over 90 minutes weekly on weeks 13-24. Patients then may undergo radiotherapy followed by trastuzumab IV over 30 minutes weekly on weeks 29-69 if they did not receive radiotherapy or on weeks 36-76 if they did receive radiotherapy.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 125 patients (100 in the neoadjuvant group and 25 in the adjuvant group) will be accrued for this study within 5 years.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed stage IIB, IIIA, IIIB, IIIC, or previously untreated stage IV primary carcinoma of the breast

  * Fine needle aspiration, core needle biopsy, or incisional biopsy allowed
  * No excisional biopsy
  * Any of the following:

    * Tumor size 2, Nodes 1 (T2N1) or tumor size 3 nodes 0 (T3N0)
    * Any T with N2 (including axillary lymph nodes matted to one another) or N3
    * Any T4, including inflammatory breast cancer
    * Adjuvant patients with at least 4 positive lymph nodes and HER-2 overexpressing tumor
    * Supraclavicular or infraclavicular positive lymph nodes without distant metastases
    * Distant metastases with measurable disease in breast or lymph nodes
* Synchronous bilateral primary breast cancer allowed if the more serious cancer meets entry criteria
* Measurable or evaluable disease

PATIENT CHARACTERISTICS:

Age: Not specified

Sex: Female

Menopausal status: Not specified

Performance status: Not specified

Life expectancy: Not specified

Hematopoietic:

White cell count > 3000 / mm3 Platelet count > 100,000 / mm3

Hemoglobin > 9 mg / dl Bilirubin < 1.5 x normal Creatinine < 1.5 x normal left ventricular ejection fraction (LVEF) normal by resting nuclear ventriculogram Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

Exclusions

Prior malignancies except:

Effectively treated squamous cell or basal cell skin cancer Carcinoma in situ of the cervix that has been curatively treated by surgery alone Nonbreast malignancy from which patient has been disease-free for 5 years and is at low risk of recurrence

Ages: 1 Year to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 1998-12; Primary Completion 2012-03 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Carey, MD, Study Chair — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trial summary from the NIH — http://grantome.com/grant/NIH/M01-RR000046-44-1159
- See also: results published in Clinical Breast Cancer — http://dx.doi.org/10.3816/CBC.2006.n.035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from University of North Carolina (UNC) at Chapel Hill and Wake Forest University School of Medicine.
Pre-assignment Details: 85 patients consented to treatment. 3 patients were consented but not treated.
Groups:
- Experimental: Herceptin With or Without Radiation: Patients will receive Adriamycin/Cytoxan (4AC) followed by Taxol plus weekly Herceptin either neo-adjuvantly or adjuvantly. Eligible patients will go on to radiation then all patients will receive additional Herceptin every three weeks for 40 weeks.
- Experimental: Non-Herceptin With or Without Radiation: Patients with high-risk human epidermal growth factor receptor 2 (HER-2) non-overexpressing tumors and those whose tumors overexpress the protein but who refuse or are ineligible for Herceptin® will be treated with conventional 4AC followed by Taxol® without Herceptin®. This will be followed by surgery then either radiation or no radiation.
Period: Overall Study
Arm/Group | Experimental: Herceptin With or Without Radiation | Experimental: Non-Herceptin With or Without Radiation
Started | 52 | 30
Completed | 52 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Non-Herceptin With or Without Radiation: Patients with high-risk human epidermal growth factor receptor 2 (HER-2) non-overexpressing tumors and those whose tumors overexpress the protein but who refuse or are ineligible for Herceptin® will be treated with conventional Adriamycin/Cytoxan (4AC) followed by Taxol® without Herceptin®. This will be followed by surgery then either radiation or no radiation.
- Total: Total of all reporting groups
Arm/Group | Experimental: Herceptin With or Without Radiation | Experimental: Non-Herceptin With or Without Radiation | Total
Number analyzed (Participants) | 52 | 30 | 82
Age, Continuous [Median (Full Range); unit: years] | 48 [24 to 69] | 48 [30 to 70] | 48 [24 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 30 | 82
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 7 | 23
  White | 35 | 21 | 56
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 52 | 30 | 82
Type of Therapy [Count of Participants; unit: Participants] — Neoadjuvant Patients: Eligible will receive four cycles of conventional dose 4AC (doxorubicin at 60 mg/m2, Cyclophosphamide at 600 mg/m2). Patients will then receive 12 weeks of weekly Taxol® (90 mg/m2) plus Herceptin® followed by surgery.
  Adjuvant Patients:
  patients will undergo surgery followed by four cycles of conventional dose 4AC (doxorubicin at 60 mg/m2, Cyclophosphamide at 600 mg/m2). Patients will then receive 12 weeks of weekly Taxol® (90 mg/m2) plus Herceptin® ( 4 mg/kg load week 1; 2 mg/kg weekly thereafter).
  Participants
    Neoadjuvant | 37 | 30 | 67
    Adjuvant | 15 | 0 | 15
Estrogen Receptor Status [Count of Participants; unit: Participants] — Fluorescence in situ hybridization (FISH) is a test that "maps" the genetic material in a person's cells. This test can be used to visualize specific genes or portions of genes. FISH testing is done on breast cancer tissue removed during biopsy to see if the cells have extra copies of the human epidermal growth factor receptor 2 (HER2) gene. The more copies of the HER2 gene that are present, the more HER2 receptors the cells have. These HER2 receptors receive signals that stimulate the growth of breast cancer cells.
  Participants
    +1 | 0 | 9 | 9
    +2 | 6 | 3 | 9
    +3 | 45 | 3 | 48
    0 | 0 | 4 | 4
    fluorescence in-situ hybridization (FISH) Negative | 0 | 11 | 11
    FISH + | 1 | 0 | 1
Clinical Stage [Count of Participants; unit: Participants] — Tumor grade is the description of a tumor based on how abnormal the tumor cells and the tumor tissue look under a microscope. It is an indicator of how quickly a tumor is likely to grow and spread. The grading system is as follows: grade I - cancer cells that resemble normal cells and aren't growing rapidly. grade II - cancer cells that don't look like normal cells and are growing faster than normal cells. grade III - cancer cells that look abnormal and may grow or spread more aggressively. Grade IV- They tend to grow quicker, spread more often and have a worse prognosis.
  Participants
    IIB | 6 | 9 | 15
    IIIA | 20 | 12 | 32
    IIIB | 8 | 6 | 14
    IIIC | 8 | 0 | 8
    IV | 10 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Toxicity of Weekly Taxol Given With Weekly Herceptin When Delivered Immediately Following Four Cycles of Standard Dose AC.
Description: Doxorubicin + cyclophosphamide in combination with paclitaxel and trastuzumab (AC-TP) Associated Systolic Dysfunction. Systolic function was measured by the ventricular ejection fraction (LVEF). LVEF is a measurement in determining how well your heart is pumping out blood and in diagnosing and tracking heart failure.
Time Frame: 78 weeks (1.5 years)
Population: LVEF data during AC-TP are complete on 50 patients. 2 are incomplete because of withdrawal (1) and progressive disease (1). 43 of the 52 patients underwent LVEF determination at 1.5 years.
Measure: Count of Participants; unit: Participants
Groups:
- Herceptin Regimen After AC: Patients in the adjuvant and neoadjuvant groups after receiving [AC-TP] Chemotherapy (doxorubicin & cyclophosphamide).
- Herceptin Regimen After TP: Patients in the adjuvant and neoadjuvant groups after receiving chemotherapy and Taxol + Herceptin.
- Herceptin Regimen at 1.5 Years: Patients in the adjuvant and neoadjuvant groups.
- Herceptin Regimen: Worst per-patient toxicity: represents the number of patients who had cardiac toxicity at any time during the study regardless of subsequent recovery of function.
Arm/Group | Herceptin Regimen After AC | Herceptin Regimen After TP | Herceptin Regimen at 1.5 Years | Herceptin Regimen
Number analyzed (Participants) | 52 | 50 | 43 | 52
Participants
  Asymptomatic LVEF < 50% | 1 | 8 | 3 | 11
  Congestive Heart Failure | 0 | 1 | 1 | 2

2. Secondary Outcome: Overall Response
Description: Measured by the Overall Response. Response: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 78 weeks (1.5 years)
Population: Protocol specifies that Response will be examined in patients who were treated neoadjuvantly. Because of this, only patients treated with Herceptin neoadjuvantly and non-Herceptin patients were included in this analysis. One patient was found unevaluable in the AC-P group and was not included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Treated Neoadjuvantly With AC-TP: Patients who were given [AC-TP] Chemotherapy (doxorubicin & cyclophosphamide) followed by paclitaxel + herceptin followed by surgery followed by radiation or no radiation followed by herceptin.
- Patients Treated With AC-P (Without Herceptin): Patients treated with AC chemotherapy followed by Taxol followed by surgery followed by radiation (or no radiation)
Arm/Group | Patients Treated Neoadjuvantly With AC-TP | Patients Treated With AC-P (Without Herceptin)
Number analyzed (Participants) | 37 | 29
Participants | 32 | 24

3. Secondary Outcome: Disease-free Survival (DFS) in Patients Receiving and Not Receiving Herceptin®.
Description: Percent of patients receiving and not receiving Herceptin who are alive and disease-free at 5 years.
Time Frame: 5 years
Measure: Number; unit: percentage of patients
Groups:
- Experimental: Herceptin With or Without Radiation: Patients who were given [AC-TP] Chemotherapy (doxorubicin & cyclophosphamide) followed by paclitaxel + herceptin in both the neoadjuvant and the adjuvant groups.
- Experimental: Non-Herceptin With or Without Radiation: Patients treated with AC chemotherapy followed by Taxol followed by surgery followed by radiation (or no radiation)
Arm/Group | Experimental: Herceptin With or Without Radiation | Experimental: Non-Herceptin With or Without Radiation
Number analyzed (Participants) | 52 | 30
percentage of patients | 69 | 60

ADVERSE EVENTS:
Time Frame: Patients were followed every 3 weeks for 74 weeks
Groups:
- Chemotherapy + Herceptin: Patients will receive Adriamycin/Cytoxan (4AC) followed by Taxol plus weekly Herceptin either neo-adjuvantly or adjuvantly. Eligible patients will go on to radiation then all patients will receive additional Herceptin every three weeks for 40 weeks.
- Control: Non-Herceptin: Patients with high-risk HER-2 non-overexpressing tumors and those whose tumors overexpress the protein but who refuse or are ineligible for Herceptin® will be treated with conventional 4AC followed by Taxol® without Herceptin®. This will be followed by surgery then either radiation or no radiation.
Arm/Group | Chemotherapy + Herceptin | Control: Non-Herceptin
All-Cause Mortality (participants affected / at risk) | 15/52 | 13/30
Serious Adverse Events (participants affected / at risk) | 7/52 | 1/30
Other Adverse Events (participants affected / at risk) | 51/52 | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + Herceptin (N=52) | Control: Non-Herceptin (N=30)
Dizziness (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Blood and lymphatic system disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0 — Transient ischemic attack
Peripheral neuropathy (Nervous system disorders) | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + Herceptin (N=52) | Control: Non-Herceptin (N=30)
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Alanine aminotransferase increased (Investigations) | 9 | 1
Alkaline phosphatase (Investigations) | 2 | 0
Allergic reaction (Immune system disorders) | 7 | 0
Anemia with transfusion (Blood and lymphatic system disorders) | 3 | 0
Anemia without transfusion (Blood and lymphatic system disorders) | 22 | 3
Anorexia (Metabolism and nutrition disorders) | 4 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 1
Aspartate aminotransferase increased (Investigations) | 7 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest pain (General disorders) | 6 | 1
Chills (General disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 8 | 0
Cystitis (Renal and urinary disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 20 | 2
Dizziness (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 5 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 | 2
Edema (General disorders) | 8 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 6 | 1
Fatigue (General disorders) | 26 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Fever (General disorders) | 2 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 2 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 0
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 8 | 1
Hot flashes (Vascular disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 4 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Infection - Other (Specify, __) (Infections and infestations) | 0 | 1
Infection w/o neutropenia (General disorders) | 5 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Insomnia (Psychiatric disorders) | 13 | 1
Kidney infection (Infections and infestations) | 1 | 0
Lymphedema (Vascular disorders) | 2 | 0
Mood Alteration (Psychiatric disorders) | 2 | 0
Mucositis (Gastrointestinal disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 23 | 20
Nail loss (Skin and subcutaneous tissue disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 8 | 0
Neuropathy (Nervous system disorders) | 39 | 22
Neutropenia w/ fever (Blood and lymphatic system disorders) | 3 | 2
Neutropenia w/o fever (General disorders) | 26 | 17
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
palpitations (Cardiac disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 3 | 0
Rectal fistula (Gastrointestinal disorders) | 1 | 0
Renal - Other (Specify) (Renal and urinary disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
Transient ischemic attack (Nervous system disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Weight Gain (Investigations) | 1 | 0
Weight Loss (Investigations) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days